CLINICAL TRIAL: NCT05562986
Title: Clinical and Biochemical Evaluation Oral Irrigator Effectiveness in Patients Under Orthodontic Treatment
Brief Title: Impacts of Oral Irrigation in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Burcu Ozkan Cetinkaya, Professor in Periodontology, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B.30.2.ODM.0.20.08/1352-1377
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Oral Hygiene; Orthodontics; Periodontal Diseases
Keywords: Cytokine(s); Matrix metalloproteinase(s); Orthodontics; Oral hygiene
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Thirty patients were randomly divided into two equal groups; patients using OI in addition to manuel brushing (OI-group), patients using IB in addition to manual brushing (IB-group). Study was planned as randomized, single-blind, parallel-design. Periodontal indexes were recorded clinically and interleukin (IL)-1β, IL-10, matrix metalloproteinase (MMP)-1, MMP-8 levels in gingival crevicular fluid were evaluated biochemically. After baseline examinations [Silness-Löe plaque index(PI), Löe-Silness gingival index(GI), probing pocket depth(PPD), clinical attachment level(CAL), bleeding on probing(BOP)], initial periodontal therapy was completed using full-mouth disinfection method. The data was collected in the baseline, 2nd, 4th and 8th weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral irrigator group (Experimental): Fifteen patients using toothbrush and oral irrigator (Aquapick, AQ-300, Aquapick Co, Ltd, Korea). All patients were told to use Modified Bass method of tooth brushing technique. PI, GI, PPD and CAL values were measured with William's probe (Hu-Fried, Chicago, IL, A.B.D) around the teeth. All clinical parameters were evaluated on each of the six regions of the teeth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual). GCF (gingival crevicular fluid) samples was collected one day after the clinical examination from buccal aspects of the mesial and distal surfaces at the interproximal sites for the evaluation of interleukin (IL)-1β, IL-10, matrix metalloproteinase (MMP)-1, MMP-8 mediators. Following the initial clinical records, all patients were performed full mouth instrumentation and described oral hygiene procedure according to their groups.
  Interventions: Diagnostic Test: GCF (gingival crevicular fluid) collection
- Interdental brush group (Experimental): Fifteen patients using toothbrush and interdental brush. All patients were told to use Modified Bass method of tooth brushing technique. PI, GI, PPD and CAL values were measured with William's probe (Hu-Fried, Chicago, IL, A.B.D) around the teeth. All clinical parameters were evaluated on each of the six regions of the teeth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual). GCF (gingival crevicular fluid) samples was collected one day after the clinical examination from buccal aspects of the mesial and distal surfaces at the interproximal sites for the evaluation of interleukin (IL)-1β, IL-10, matrix metalloproteinase (MMP)-1, MMP-8 mediators. Following the initial clinical records, all patients were performed full mouth instrumentation and described oral hygiene procedure according to their groups.
  Interventions: Diagnostic Test: GCF (gingival crevicular fluid) collection

INTERVENTIONS:
Diagnostic Test: GCF (gingival crevicular fluid) collection — Prior to GCF (gingival crevicular fluid) sampling, supragingival plaque was removed by sterile curets and, after air drying, the surfaces were isolated by cotton rolls. Filter paper strips (periopaper, proflow Inc., Amityville, NewYork, USA) were placed in sulcus for 30s. Care was taken not to avoid mechanical trauma and strips contaminated with blood or saliva were discarded. The absorbed GCF volume was estimated by a calibrated instrument (periotron 8000, proflow Inc., Amityville, NY, USA). Then, the strips were sealed into sterile tubes before freezing at -80 0C. The readings were converted to an actual volume (μl) by reference to the standard curve.

SUMMARY:
The present study aimed to investigate clinically the cleaning effectiveness of different treatment modalities, that is, oral irrigator or interdental brush usage addition to routine brushing and examine interleukin (IL)-1β, IL-10, matrix metalloproteinase (MMP)-1, MMP-8 levels in gingival crevicular fluid of orthodontic patients. The null hypothesis was that oral irrigators would be effective compared to interdental brush in the oral care of individuals who are orthodontic patients.

DETAILED DESCRIPTION:
The aim of this study is to compare the effectiveness of oral irrigator (OI) with interdental brush (IB) clinically and biochemically in orthodontic patients.

Thirty patients were randomly divided into two equal groups; patients using OI in addition to manuel brushing (OI-group), patients using IB in addition to manual brushing (IB-group). Study was planned as randomized, single-blind, parallel-design. Periodontal indexes were recorded clinically and interleukin (IL)-1β, IL-10, matrix metalloproteinase (MMP)-1, MMP-8 levels in gingival crevicular fluid were evaluated biochemically. After baseline examinations [Silness-Löe plaque index(PI), Löe-Silness gingival index(GI), probing pocket depth(PPD), clinical attachment level(CAL), bleeding on probing(BOP)], initial periodontal therapy was completed using full-mouth disinfection method. The data was collected in the baseline, 2nd, 4th and 8th weeks.

The hypothesis of our study is that oral irrigators may be effective in oral care of orthodontic patients because of the ease of use.

ELIGIBILITY:
Inclusion Criteria:

* Being over 12 years old.
* Having at least 20 permanent teeth with bands or brackets.
* Finished phase I periodontal treatment.
* Bleeding below 10% during probing.
* No pocket depth of more than 5 mm.
* Not receiving any treatment other than orthodontic treatment during the study.
* Absence of removable or fixed prosthetic restorations.
* Absence of any systemic disease (hepatic, renal, hematologic, cardiovascular).
* Agreeing not to use any non-study mouthwash throughout the study.

Exclusion Criteria:

* Performing poor cooperation.
* Having diseases associated with bacteriemia.
* Used antibiotics and anti-inflammatory drugs for any purpose for a long time.
* Having diabetes.
* Smoking habits.
* Having a physical or mental problem that affects manual dexterity.
* Using medication that could affect gingival health (such as dilantin, calcium channel blocker, cyclosporine, and anticoagulant).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
GCF (gingival crevicular fluid) level of IL-1β as a marker of gingival inflammation | through study completion, an average of 1 year
  Elevated levels of IL-1β in GCF have been associated with the destructive changes that occur in the inflamed human gingiva, is a proinflammatory cytokine.
GCF (gingival crevicular fluid) level of IL-10 as a marker of gingival inflammation | through study completion, an average of 1 year
  IL-10 plays an important role as a stop signal in suppressing the immune and inflammatory response by being released from periodontal tissues, thus trying to limit the spread and severity of the disease. It is an anti-inflammatory cytokine. It is reported that the level of GCF IL-10 is increased in inflamed areas.
GCF (gingival crevicular fluid) level of MMP-1 as a marker of gingival inflammation | through study completion, an average of 1 year
  One of the MMPs, MMP-1, is generally expressed by fibroblasts, endothelial cells, keratinocytes, monocytes/macrophages, chondrocytes, and osteoblasts, and is a key regulator in connective tissue remodeling. In addition to gingivitis, there is a significant increase in MMP-1 levels in the GCF during the active periods of periodontitis.
GCF (gingival crevicular fluid) level of MMP-8 as a marker of gingival inflammation | through study completion, an average of 1 year
  High concentration of MMP-8 is associated with tissue destruction and severity of periodontal disease. It is known to be secreted from inflammatory cells such as neutrophils and macrophages.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu OZKAN CETINKAYA, Prof, Study Director — Ondokuzmayis University, Faculty of Dentistry, Department of Periodontology, Samsun, Turkey.; Esma SAHIN, Dr, Principal Investigator — Erzurum Public Oral Health Center, Erzurum, Turkey.; Bahattin AVCI, Prof, Study Chair — Ondokuzmayis University, Faculty of Medicine Department of Biochemistry, Samsun, Turkey.; Selma ELEKDAG TURK, Prof, Study Chair — Ondokuzmayis University, Faculty of Dentistry, Department of Orthodontics, Samsun, Turkey.
Locations (1):
- Ondokuz Mayıs University, Faculty of Dentistry, Department of Periodontology, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No